# Official title: Early Childhood Outside (ECO) Early Childhood Educator (ECE) Tool - Randomized Controlled Trial Study

NCT number: NCT04624932

Document date: October 10, 2020

Document type: Cover letter form (i.e., consent form)



# Early Childhood Outside: Early Childhood Educator Tool Randomized Controlled Trial (RCT) Study

#### Cover Letter

## Title of Study:

Early Childhood Outside: Early Childhood Educator Tool Randomized Controlled Trial (RCT) Study

# **Principal Investigator**

**Dr. Mariana Brussoni**, Department of Pediatrics, University of British Columbia; BC Children's Hospital Research Institute.

Email: mbrussoni@bcchr.ca; Tel: 604-875-3712

## **Sponsor**

This study is funded by the Lawson Foundation.

#### **Purpose**

Outdoor play is important for children as it can promote healthy social and physical development, emotional wellbeing, self-confidence, risk management and overall physical activity. However, opportunities for outdoor play have been decreasing across generations due to perceptions that it is dangerous and unnecessary. To help early childhood educators learn the importance of outdoor play, and develop strategies to give children at their centre more opportunities for outdoor play, we developed an online educational tool. The aim of the current study is to test the effectiveness of this online tool in reframing early childhood educators' perceptions of outdoor play and changing their service delivery to give children at their centre more opportunities for outdoor play.

You are being invited to take part in this study because you are 19 years old or older, currently working as an early childhood educator and/or administrator in Canada, and can speak, read and understand English.

# **Study Procedures**

If you agree to participate, you will be randomly assigned to one of the two groups: 1) Control group, or, 2) Intervention group. Neither the researchers, nor you will know in advance which group you will be assigned to. There is a ½ chance that you are assigned to any group. After you are randomized to one of the two groups, you will be asked to complete demographic and survey questionnaires. Demographic questions

are asked to understand general background information about yourself (e.g., sex, age) and your ECE centre (e.g., approximately how many staff are at your centre). These questionnaires can take up to 20 minutes to complete.

If you are assigned to the Control group, you will be provided with generic information about children's outdoor play, which can take up to 20 minutes to read. Then, you will be invited to set a goal that could help you give children at your centre more opportunities for outdoor play.

If you are assigned to the Intervention group, you will be automatically taken to our online tool. The online tool is to reframe your perceptions of outdoor play and change your service delivery in promoting children's outdoor play at your centre. It includes a series of interactive video scenarios where you can make choices, which will result in different endings for each scenario. This can take up to 100 minutes to complete. Then you will be invited to set a goal that could help you give children at your centre more opportunities for outdoor play. If you are assigned to the Control group, you will have access to the online tool upon completion of your participation in the current study.

After 1 week, you will receive an email from us to invite you to complete the same survey questionnaire for the second time. We will also follow up whether you had accomplished your goal. This round of survey questionnaires can take up to 10 minutes.

After 3 months, you will receive another email from us to invite you to complete the same survey questionnaire for the final time. We will also follow up whether you had accomplished your goal. This round of survey questionnaires can take up to 10 minutes.

Study procedure and time commitment are as below:

| Enrollment | |
|----------------------------------------|---------------------|
| Baseline survey | |
| [up to 20 minutes] | |
| Randomization to one of the two groups | |
| Control | Intervention |
| Generic information | Our online tool |
| [up to 20 minutes] | [up to 100 minutes] |
| Honorarium: \$30 | Honorarium: \$30 |
| 1 week after baseline | |
| Follow-up survey | |
| [up to 10 minutes] | |
| Honorarium: \$25 | |
| 3 months after baseline | |
| Follow-up survey | |
| [up to 10 minutes] | |
| Honorarium: \$25 | |

#### **Potential Risks**

No risks are expected as a result of participating in this study. Nonetheless, if you feel any distress during the study, or simply no longer wish to participate, you can withdraw from the study at any time without any penalty.

# **Potential Benefits**

While there may not be any direct benefit from participating in this study, potential benefits can result from learning the benefits of outdoor play for children, which can be applied in your own child care practice.

# **Confidentiality**

Your confidentiality will be respected. You will be assigned a unique study number as a participant in this study. This number will not include any personal information that could identify you. Research records and data that can indirectly identifying you (e.g., email address) may, nonetheless, be inspected in the presence of the Principal Investigator by representatives of the Lawson Foundation, Health Canada, and University of British Columbia Research Ethics Board for the purpose of monitoring the research. No information or records that disclose your identity will be published without your consent, nor will any information or records that disclose your identity be removed or released without your consent unless required by law.

Your rights to privacy are legally protected by federal and provincial laws that require safeguards to ensure that your privacy is respected. You also have the legal right of access to the information about you that has been collected for this study, and an opportunity to correct any errors in this information, if needed. Further details about these laws are available on request to your study researcher.

Your data will be stored in a password protected folder in a secured network at the BC Children's Hospital Research and Google Analytics for 5 years post completion of study. Only the research team associated with the study will have access to them for the purpose of data processing, cleaning and analysis. After 5 years post completion of study, these will be destroyed (i.e., permanently deleted) wherever possible.

# Remuneration/Compensation

To acknowledge your time and contribution to the study, you will receive \$30 upon completion of the baseline survey and then \$25 for each follow-up survey you complete (1 week and 3 months after baseline), a total of \$80. You will receive your honoraria via e-Interact using your email address.

## Contact for information about the study

If you have any questions or concerns about what we are asking of you, please contact Dr. Mariana Brussoni at <a href="mailto:mbrussoni@bcchr.ca">mbrussoni@bcchr.ca</a> or 604-875-3712, or Christina Han, research coordinator at <a href="mailto:chan@bcchr.ca">chan@bcchr.ca</a> or 604-875-2000 ext. 2433.

# Contact for concerns about the rights of research subjects

If you have any concerns or complaints about your rights as a research participant and/or your experiences while participating in this study, contact the Research Participant Complaint Line in the University of British Columbia Office of Research Ethics by e-mail at RSIL@ors.ubc.ca or by phone at 604-822-8598 (Toll Free: 1-877-822-8598). Please reference the study number (H19-03644) when contacting the Complaint Line so the staff can better assist you.

## Consent

By completing the questionnaire, you are consenting to participate in this research.

Providing consent assumes that:

- The study has been fully explained to you and all of your questions have been answered;
- You understand the requirements of participating in this study which could include up to 140 minutes in total:
- You understand that you have the right not to take part in the study and the right to stop at any time;
- You have been informed of the potential risks and benefits of the study; and,
- You understand that your information collected in this study (except for your email address) will be used for the current and potential future data analyses.

Would you like to be contacted for future similar studies? If yes, we'll contact you via email you share in the survey.

- o Yes
- o No

Please save a copy of this document for your records.